CLINICAL TRIAL: NCT05303077
Title: The Effect of a New Newborn Formula Over the Corporal Composition: a Randomized Multicentric Clinical Trial
Brief Title: Study of the Effects of a New Infant Formula Supplemented With a Probiotic Over the Corporal Composition of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alter Farmacia, S.A. (Industry)
Collaborators: Fundación Teófilo Hernando, Spain (Other); Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: INNOVA 2020
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Infant formula, body composition, safety
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The 2 infant formula arms are blinded for the participant, investigator and data analyst. The 3rd arm is an open control group conformed by breastfeed infants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Infant Formula (Experimental): Infant formula supplemented with omega 3 fatty acids and inactive Bifidobacteria
  Interventions: Dietary Supplement: Nutribén Innova® 1
- Infant Formula (Active Comparator): Infant formula
  Interventions: Dietary Supplement: Nutribén®
- Breastfeed Active comparator (Active Comparator): Infants who are breastfed
  Interventions: Dietary Supplement: Breastfeed

INTERVENTIONS:
Dietary Supplement: Nutribén Innova® 1 — Infants are fed solely with infant formula supplemented with an inactive probiotic and omega 3 fatty acids over the first 6 months of their life, from then on the infants are fed with the study formula and the usual supplementary food, recommended to the baby's
  Arms: Study Infant Formula
Dietary Supplement: Nutribén® — Infants are fed solely with infant formula over the first 6 months of their life, from then on the infants are fed with the study formula and the usual supplementary food, recommended to the baby's age.
  Arms: Infant Formula
Dietary Supplement: Breastfeed — Infants are breastfeeding solely over the first 6 months of their life, from then on the infants are fed as recommended by their caregiver, as if they are not participating in a research study.
  Arms: Breastfeed Active comparator

SUMMARY:
This is a multicentric, randomized, blinded, controlled trial to study the effects of a new infant formula on the changes in the newborn body composition over time: weight gain, anthropometric data, incidence of infections, digestive tolerance (flatulence, vomiting and regurgitation), feces (consistency and frequency), behavior (restlessness, colic, nocturnal awakenings), count of probiotic strains of the intestinal microbiota in feces, safety and tolerability of the investigational products (measured as number, frequency and severity of adverse events in all branches of the study)

ELIGIBILITY:
Inclusion Criteria:

* Healthy children. Both sex.
* Full term infants (between 37 and 42 weeks of pregnancy).
* Birth weight between 2500 g- 4500 g.
* Single birth babies.
* BMI of the mothers before the pregnancy between 19 y 30 kg/m2.

Exclusion Criteria:

* Body weight lower than the 5th percentile for their gestational age.
* Cow's milk protein allergy and/or lactose allergy.
* Administration of antibiotics 7 days prior inclusion.
* Congenital disease or malformation that may affect the infant growth rate.

Population Description: The study population are newborns selected from primary care clinics in Spain.

Sampling Method: Not applicable

* Metabolic disease or disorders.
* Significant prenatal disease and/or serious postnatal disease before recruitment.
* Underage parents.
* Diabetic mother.
* Born from a drug abuse mother (who use abuse drugs during pregnancy).
* Parents cannot comply with study procedures.
* Subject included or that have been included in other clinical trial since his/her birth day.

Ages: 15 Days to 25 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Weight gain at 6 months | 6 months after the beginning of the study
  Measure of weight gain by grams/day between the first visit and month 6

SECONDARY OUTCOMES:
weight at 21 days, 2, 4, 6 and 12 months | 21 days, 2, 4, 6 and 12 months
  Measure of weight gain by grams
Length gain | 21 days, 2, 4, 6 and 12 months
  Measure of the infant's length gain over time in cms
Head circumference gain | 21 days, 2, 4, 6 and 12 months
  Measure of the increase of the head circumference over time in cms
Tricipital Skin fold development | 4, 6 and 12 months
  Measurement of the development of tricipital skin fold, in cms, measured using a skinfold caliper
Subscapular skin fold develompent | 4, 6 and 12 months
  Measurement of the development of subscapular skin fold, in cms, measured using a skinfold caliper
Mean arm circumference | 4, 6 and 12 months
  Measure of arm circumference over time in cms.
Feces features consistency | 21 days, 2, 4, 6 and 12 months
  Description of the consistency of baby's feces features, according to their parent's perception, on a qualitative scale: soft, hard, liquid, normal, semiliquid, pasty. The analysis includes the number of feces in each group and the overall frequency by study arm and visit.
Feces features number of bowel movements | 21 days, 2, 4, 6 and 12 months
  Number of bowel movements per day sorted by study group
Digestive tolerance | 4, 6 and 12 months
  The digestive tolerance will be assessed as adequate, constipation, flatulence, vomit or other distresses, which are a heterogeneous group that includes various affections as diarrhea, abdominal pain, irritability, constipation, regurgitation or colic. The analysis includes the overall number and the frequency sorted by study arm.
Infant's behavior | 4, 6 and 12 months
  Qualitative variable. The infant's behavior is classified as either good or altered. The total number and the relative frequency by group are included in the analysis.
intestinal microbiota | 4, 6 and 12 months
  Analysis of the evolution of the intestinal microbiota of the children over the study. The richness and diversity of the microbiota are analyzed and compared between the study groups.
Evolution of calprotectin levels in feces | 21 days, 2, 6 and 12 months
  Measurement of the evolution of calprotectin levels in feces over time
Evolution of IgA levels in feces | 21 days, 2, 6 and 12 months
  Measurement of the evolution of IgA levels in feces over time
Evolution lactic acid levels in feces | 21 days, 2, 6 and 12 months
  Measurement of the evolution of lactic acid levels in feces over time
Evolution of short-chain fatty acid levels in feces | 21 days, 2, 6 and 12 months
  Measurement of the evolution of short-chain fatty acid levels in feces over time
Morbility | over a year
  Analysis of the number and frequency of all adverse events registered during the study by feeding group
Products Tolerability | over a year
  Quantitative variable. The tolerability of the products is assessed as adequate, good, very good, unsatisfactory. The analysis includes the overall number y and the relative frequency by group.
Overall rate of the products | 2, 4, 6 and 12 months
  Quantitative variable. The parents' subjective rate of the products. The assessment can be, acceptable, good, very good, satisfactory or not satisfactory.

CONTACTS AND LOCATIONS:
Locations (21):
- Spain (21):
  - Cap Montclar, Barcelona
  - Cap Nova Lloreda, Barcelona
  - Cap Sant Ildefons, Barcelona
  - Consulta Dr. Xavier Riopedre, Barcelona
  - Consulta Carlos Nuñez de Prado Aparicio, Madrid
  - Consultorio Arroyomolinos (Cs Parque Coimbra), Madrid
  - Cs Alcalde Bartolomé Gonzalez Móstoles, Madrid
  - Cs Conde de Barcelona, Madrid
  - Cs Dr Luengo Rodríguez, Madrid
  - Cs Infante Don Luis de Borbón, Madrid
  - Cs La Rivota, Madrid
  - Cs Las Américas, Madrid
  - Cs Miguel Servet, Madrid
  - Cs Parque Loranca, Madrid
  - Cs Presentación Sabio, Madrid
  - Cs Valle de La Oliva, Madrid
  - Clínica Dr Aguilar-Dr Sacristán, Seville
  - Consultas Externas Hospital Privado Santa Ángela de La Cruz, Seville
  - Cs Amante Laffón, Seville
  - Cs Utrera Norte, Seville
  - Ihp Bellavista, Seville